CLINICAL TRIAL: NCT03036540
Title: Symptomatic and Asymptomatic Thrombosis in Midline Catheter
Brief Title: Upper Limb Thrombosis Associated With Midline Catheter
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, jiri charvat, prof.MD, PhD, University Hospital, Motol
Other Study IDs: UHMotol6022
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Venous Thrombosis Deep (Limbs)
Keywords: upper limb thrombosis, midline catheter
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: application in midline catheter — The routine insertion of midline catheter for the patients admitted in hospital who needs peripheral venous approach for the period more than 5 days or with the insufficient peripheral veins system

SUMMARY:
The patients admitted in hospital who had midline catheter inserted in upper limb are followed-up for the presence of complications related to catheter introductions. The symptoms and signs of upper limb thrombosis are recorded. The diagnosis is confirmed by sonography examination. In the selected group of asymptomatic patients sonography examination is done 8 to 10 days after cathether insertion in order to detect the incidence of the asymptomatic thrombosis

DETAILED DESCRIPTION:
The patients admitted in hospital who had midline catheter inserted in upper limb are followed-up for the presence of complications related to catheter introductions. The symptoms and signs of upper limb thrombosis are recorded. The diagnosis is confirmed by sonography examination. The age, gender, principal diagnosis, the vein were midline catheter is inserted and number of vein punctures for catheter insertion are recorded. Afterward the patients are treated in the ward and the possible complications are recorded. The main concern is about the incidence of upper limb thrombosis. All the complications are recorded as well as date when they has appeared. The statistical analysis is done in order to evaluate the incidence of upper limb symptomatic thrombosis, the duration since insertion to thrombosis manifestation ańad its associations with age, gender, principal diagnosis, selected vein, its size and number of punctures is analysed.

In the selected group of the asymptomatic patients 8 to 10 days after midline insertion upper limb sonography is done in order to detect the presence of the asymptomatic upper limb thrombosis and the same type of analysis as for symptomatic thrombosis is undertaken.

ELIGIBILITY:
Inclusion Criteria:

* The patients admitted to University Hospital suffering from disease when venous access is required for period longer than 5 days or with insufficient peripheral venous access

Exclusion Criteria:

The patients who need another type of venous access, e.g. central venous access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients admitted to University Hospital suffering from disease when venous access is required for period longer than 5 days or with insufficient peripheral venous access
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
The symptomatic and asymptomatic upper limb thrombosis in the patients with midline catheter | admitted patients in hospital during one year with midline catheter insertion
  The detection of the incidence of upper limb thrombosis and definition of the associated factors

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Charvat, MD,PhD, Study Chair — University Hospital, Motol
Locations (1):
- University hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No
The patients with the inseertion of midline catheter during admission in hospital are followed-up for the possible complications including symptoms and signs of symptomatic and asymptomatic upper limb thrombosis using sonography examinations